CLINICAL TRIAL: NCT03064945
Title: A Randomized, Controlled, Multi-Center, CROSSOVER, Prospective, Double-blind Clinical Study to Assess the Effectiveness and Safety of Livia® Transcutaneous Electrical Nerve Stimulation (TENS) in Women Suffering From Primary Dysmenorrhea
Brief Title: The Effectiveness and Safety of LIVIA® Transcutaneous Electrical Nerve Stimulation (TENS) in Women Suffering From Primary Dysmenorrhea.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: iPulse Medical Ltd. (Livia) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIVIA-01
Record Dates: First submitted 2017-02-22; First posted 2017-02-27 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2017-05

CONDITIONS: Dysmenorrhea
Keywords: Livia TENS; safety and efficacy; menstruating women
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Shame device (Sham Comparator)
  Interventions: Device: Livia
- Livia® Transcutaneous Electrical Nerve Stimulation (TENS) (Experimental)
  Interventions: Device: Livia

INTERVENTIONS:
Device: Livia — Livia® Transcutaneous Electrical Nerve Stimulation (TENS) is a novel pain management device for women suffering from dysmenorrhea

SUMMARY:
This is a randomized, controlled, multi-center, single-arm, crossover, double-blind clinical study assessing the Livia Transcutaneous Electrical Nerve Stimulation (TENS) in women suffering from dysmenorrhea. The study will be conducted at community clinics. Advertisement will be used to publish and promote recruitment.

The study will include 3 visits: Screening visit and two consecutive visits each one after monthly menstrual period. Treatment will be self-administrated and during the study, the subjects will be requested to complete home diaries.

ELIGIBILITY:
Inclusion Criteria:

1. Women between the age 18 to 45 years
2. Women reporting painful menstruation during the last 3 menstrual cycles.
3. Pain VAS score of at least 60 based on previous menstrual cycle
4. Subject is willing and able to comply with the study protocol and provide written informed consent to participate in the study.
5. Subject must agree to consistently use effective contraception throughout the study. (Subject not treated with oral contraception should use any contraception other than oral).

Exclusion Criteria:

1. Participation in any other investigational study within 30 days prior and/or at the date of subject consent.
2. Woman with a significant medical condition such as: cancer, diabetes (Type I and II), irritable bowel disease IBD, immunodeficiency, autoimmune disease, etc. that in the investigator opinion, participation in the study would place the patient at an unacceptable risk.
3. Pregnant woman
4. A woman who is diagnosed with secondary dysmenorrhea associated with uterine myomas, endometriosis, adenomyosis, etc.
5. A woman who has cardiac condition with cardiac pacemakers, implanted defibrillators, or other implanted metallic or electronic devices.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study on women that suffering from painful menstruation
Enrollment: 63 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-04-25 (Actual); Study Completion 2018-04-25 (Actual)

PRIMARY OUTCOMES:
The difference between the reported Visual Analogue Scale before and after applying the device (active or sham). | 3 days before the beginning of the menstrual period and up to three days after termination of the menstrual period.
  Each participant will rank the severity of her dysmenorrhea symptoms before and after the device use on the VAS scale from 0 to 100, where 0 determines- "No pain" and 100 determines "Very painful". Then, the difference between the two measurements will be calculated.

SECONDARY OUTCOMES:
Usage of pain relievers during the menstrual period | 3 days before the beginning of the menstrual period and up to three days after termination of the menstrual period.
  Usage of pain relievers during the menstrual period as recorded in the subjects' diaries. This will be measured by the number of pain relief pills taken during the entire menstrual period
Quality of life | 3 days before the beginning of the menstrual period and up to three days after termination of the menstrual period.
  Quality of life will be assessed using the Q-LES Questionnaire. The summary score will be determined as per the questionnaire manual
The convenience of device operation | 3 days before the beginning of the menstrual period and up to three days after termination of the menstrual period.
  The convenience of device operation and usage will be determined using a series of specific questions posed to the subjects at visit 3.

OTHER OUTCOMES:
SAFETY AND TOLERABILITY ENDPOINTS | 3 days before the beginning of the menstrual period and up to three days after termination of the menstrual period.
  The safety and tolerability endpoints of this study are Adverse events (AEs) and serious adverse events (SAEs) occurring at any time during the study Duration of device use

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah, Jerusalem, Israel